CLINICAL TRIAL: NCT06462222
Title: Immune Checkpoint Inhibitor Combined With Pemetrexed Intrathecal Injection for Leptomeningeal Metastasis From Solid Tumors: a Phase I/II Study
Brief Title: Immune Checkpoint Inhibitor Combined With Pemetrexed Intrathecal Injection for Leptomeningeal Metastasis From Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPLM
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Leptomeningeal Metastasis
Keywords: Leptomeningeal metastasis; Intrathecal chemotherapy; Immune checkpoint inhibitor; Pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — toripalimab; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group (Experimental): Immune checkpoint inhibitor combined with pemetrexed
  Interventions: Drug: Toripalimab, pemetrexed

INTERVENTIONS:
Drug: Toripalimab, pemetrexed — Drug 1: Toripalimab 40 mg; Drug 2: pemetrexed 15mg. intrathecal injection therapy

SUMMARY:
This is an open-label, single-arm, phase I/II trial of immune checkpoint inhibitor combined with pemetrexed intrathecal injection for leptomeningeal metastasis from solid tumors.

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase I/II trial of immune checkpoint inhibitor combined with pemetrexed intrathecal injection for leptomeningeal metastasis from solid tumors. The primary objective was to assess recommended dose and safety based on adverse events (AEs). All participants were observed to evaluate the clinical response rate (CRR), disease control rate (DCR) and overall survival (OS). Patients underwent cerebrospinal fluid (CSF) and blood specimen collection to evaluate potential clinical, molecular, and/or immune predictors of treatment efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of solid tumors; Cerebrospinal fluid cytopathology is positive.
2. Male or female aged between 18 and 75 years; Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.
3. No history of severe nervous system disease; No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. A history of HIV or AIDS, acute or chronic hepatitis B or C infection, previous anti-PD1 therapy-induced pneumonitis, or have ongoing >Grade 2 adverse events of such therapy; or ongoing autoimmune disease that required systemic treatment in the past 2 years.
4. Patients with poor compliance or other reasons that were unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Recommended dose | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.]
  The recommended dose of intrathecal PD-1 inhibitor. The dose limiting toxicity was defined as ≥ grade 3 neurological toxicities (e.g., chemical meningitis) or other grade 4 toxicity.
Incidence of treatment-related adverse events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE). Events of grade 3-5 are defined as moderate and severe adverse events.

OTHER OUTCOMES:
Clinical response rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Progression-free survival related to leptomeningeal metastasis (LMPFS) | From date of treatment until the date of first documented leptomeningeal metastasis progression or date of death from any cause, whichever came first, assessed up to 6 months.
  LMPFS was defined as time from the start of treatment until leptomeningeal metastasis progression or death. The leptomeningeal metastasis progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.
Overall survival(OS) | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up (at least 7 months).
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huizhou Hospital, Guangzhou Medical University, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete

REFERENCES:
- [Background] Glitza Oliva IC, Ferguson SD, Bassett R Jr, Foster AP, John I, Hennegan TD, Rohlfs M, Richard J, Iqbal M, Dett T, Lacey C, Jackson N, Rodgers T, Phillips S, Duncan S, Haydu L, Lin R, Amaria RN, Wong MK, Diab A, Yee C, Patel SP, McQuade JL, Fischer GM, McCutcheon IE, O'Brien BJ, Tummala S, Debnam M, Guha-Thakurta N, Wargo JA, Carapeto FCL, Hudgens CW, Huse JT, Tetzlaff MT, Burton EM, Tawbi HA, Davies MA. Concurrent intrathecal and intravenous nivolumab in leptomeningeal disease: phase 1 trial interim results. Nat Med. 2023 Apr;29(4):898-905. doi: 10.1038/s41591-022-02170-x. Epub 2023 Mar 30. PMID 36997799
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065